CLINICAL TRIAL: NCT02105142
Title: Comparative Effectiveness of Primary Care-based Interventions for Pediatric ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nerissa Bauer, Assistant Professor, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1305011436
Record Dates: First submitted 2014-03-30; First posted 2014-04-07 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention deficit hyperactivity disorder; Interventions; Primary care; Pediatric
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Computer Decision Support (Active Comparator): ADHD Module of the Child Health Improvement through Computer Automation (CHICA) system Designed to facilitate physician adherence to clinical care guidelines for ADHD identification and chronic care management
  Interventions: Behavioral: Computer Decision Support
- ADHD Group visits (Active Comparator): Parents and children attend separate but concurrently run group visits every three months; groups are facilitated by general pediatricians
  Interventions: Behavioral: ADHD Group Visits
- ADHD Group Visits plus Online Discussion Portal (Active Comparator): Parents and children attend separate but concurrently run group visits every three months; groups are facilitated by general pediatricians. Online discussion portal access granted to parent participants and will allow parents to communicate with each other in between in-person group visits
  Interventions: Behavioral: ADHD Group Visits plus Online Discussion Portal

INTERVENTIONS:
Behavioral: ADHD Group Visits — Parents and children attend separate but concurrently run group visits every three months; groups are facilitated by general pediatricians
  Arms: ADHD Group visits
Behavioral: ADHD Group Visits plus Online Discussion Portal — Parents and children attend separate but concurrently run group visits every three months; groups are facilitated by general pediatricians. Parent participants will be granted access to the online discussion portal to allow for communication in between in-person group visits.
  Arms: ADHD Group Visits plus Online Discussion Portal
Behavioral: Computer Decision Support — ADHD Module of the Child Health Improvement through Computer Automation (CHICA) system Designed to facilitate physician adherence to clinical care guidelines for ADHD identification and chronic care management
  Arms: Computer Decision Support

SUMMARY:
Attention-deficit hyperactivity disorder (ADHD) is the most common neurobehavioral disorder of childhood, affecting approximately 8% of youth. Children with ADHD often have problems sustaining attention and completing multi-step commands and tasks of daily living, such as homework. Pediatricians are often the first physicians to identify problems with children's functioning at home and at school. However, because of limited visit time, pediatricians often struggle with managing ADHD while trying to also cover a vast array of other primary care issues. Moreover, as there is a nationwide shortage of pediatric mental health specialists and access to parenting programs is limited, a critical need exists to develop interventions that form partnerships between behavioral and mental health specialists and the primary care pediatrician. One approach is to base interventions in the pediatric clinic to ensure children have access to appropriate treatment. Thus far, only a limited number of sites have this pediatric-mental health partnership.

Health information technology (HIT) has been used to enhance primary care management of ADHD. HIT can improve pediatricians' ability not only to adhere to recommended guidelines, but also to screen for co-existing disorders and provide timely parental education. An alternative strategy might be to use group visits (GV). GV afford more time with families and allows the pediatrician to facilitate more in-depth discussions. More importantly, the group model allows parents to learn from one another, normalizes parenting expectations, and addresses shared experiences of medication side effects and other factors related to adherence. Moreover, a group visit can be conducted in a physical location, such as the pediatric clinic, or be brought into the virtual world with the aid of social media. Virtual support groups for chronic care diseases have become an increasingly popular way for a community of individuals to exchange information and offer emotional support.

Prior to the adoption of these interventions into primary care practice, investigators must know which is best. Rigorous comparative effectiveness research (CER) can help to determine this. This proposal will compare a HIT based intervention to a GV strategy, with and without the use of social media. These 3 interventions will be compared based not only on clinical measures of interest but also on parent-defined patient outcomes. Prior research has largely focused on measuring clinical outcomes such as treatment adherence and ADHD symptom reduction with little emphasis on understanding how patient-centered outcomes, such as the quality of life of families dealing with ADHD, are affected.

Building on previous work, the specific aims for this study are:

Aim 1. Compare the preliminary efficacy of three interventions to improve treatment of ADHD in the primary care setting Aim 1a) Compare the effectiveness of the three interventions on clinical measures such as parent and teacher rated ADHD symptoms and adaptive functioning Aim 1b) Compare the effectiveness of the three interventions on patient-centered outcomes such as quality of life and parental satisfaction with the intervention The three interventions will be: 1) Child Health Improvement through Computer Automation (CHICA) which is the health information technology innovation arm; 2) Group visits (GV); or 3) Group visits plus online discussion portal (GV+DP).

ELIGIBILITY:
Inclusion Criteria:

* Children 6 to 12 years of age with diagnosis of ADHD and their parents
* Children must receive medical care at participating study clinics
* Children must have diagnosis of ADHD based on parent and teacher diagnostic and statistical manual-IV rating scales
* Children can have co-existing Oppositional Defiant Disorder (ODD)

Exclusion Criteria:

* Children with co-existing diagnosis of Conduct Disorder (CD)
* Children with autism
* Children with moderate to severe mental handicap or other neurodevelopment disorder that would preclude active participation in group discussions

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in Vanderbilt ADHD Rating Scale scores | Baseline & 12 months
  ADHD symptoms as measured by parent-report and based on Diagnostic and Statistical Manual-IV diagnostic criteria.

SECONDARY OUTCOMES:
Change in scores for pediatric quality of life | Baseline & 12 months
  Quality of Life (generic core scales): 23 items, related to quality of life and child's needs in context of the family. Parent and child report.
Change in score of multidimensional scale of perceived social support scale | Baseline & 12 months
  Social Support: 12-items perceptions on support
Parental Locus of Control-Short Form | Baseline
  Locus of Control: 25-items, degree parent feels in control of child behavior
Change in scores related to adaptive functioning | Baseline & 12 months
  13 items, parent-report, measuring adaptive functioning in the home using the Home Situations Questionnaire. Responses at each separate time point will be compared to the study specific Childhood ADHD and Family Impact Scale scores for correlation.
Change in scores on Childhood ADHD & Family Impact Scale | Baseline & 12 months
  Study-specific tool, 9 items related to common challenges related to parenting based on feedback by patient advisory board

OTHER OUTCOMES:
Demographics | Baseline
  Study-specific tool,12 items capturing demographics & characteristics of participant
Satisfaction with content of group visits | Every 3 months at the end of each attended group visit
  Separate forms for parent and child feedback on group visits (5-6 items, 1 page); subjects in GV or GV-DP only
Pediatric facilitator feedback form | Every 3 months at the end of each attended group visit
  Parent ratings of communication, teaching style and preparedness of pediatric facilitator; subjects in GV or GV-DP only
Discussion portal feedback form | 12 months
  Closed and open ended questions about: if parent accessed the online discussion portal (yes/no), how often accessed (daily/weekly/monthly/never), perceived benefits of the online discussion portal, any suggestions for usefulness; subjects in GV-DP only
Adherence to ADHD Group Visit curriculum | Every month for 15 months
  Protocol checklist for each session to be completed by facilitators after each session and by study team to monitor adherence; facilitators and study team only

CONTACTS AND LOCATIONS:
Overall Officials: Nerissa S Bauer, MD, MPH, Principal Investigator — Indiana University School of Medicine
Locations (5):
- United States (5):
  - General Pediatrics Clinic Medical Service Area 1 in Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Eskenazi Health Center-Blackburn, Indianapolis, Indiana
  - Eskenazi Health Center- Forest Manor, Indianapolis, Indiana
  - Eskenazi Health Center-W. 38th Street, Indianapolis, Indiana
  - Eskenazi Health Center- Pecar, Indianapolis, Indiana

REFERENCES:
- [Background] Carroll AE, Bauer NS, Dugan TM, Anand V, Saha C, Downs SM. Use of a computerized decision aid for ADHD diagnosis: a randomized controlled trial. Pediatrics. 2013 Sep;132(3):e623-9. doi: 10.1542/peds.2013-0933. Epub 2013 Aug 19. PMID 23958768
- [Derived] Bauer NS, Sullivan PD, Szczepaniak D, Stelzner SM, Pottenger A, Ofner S, Downs SM, Carroll AE. Attention Deficit-Hyperactivity Disorder Group Visits Improve Parental Emotional Health and Perceptions of Child Behavior. J Dev Behav Pediatr. 2018 Jul/Aug;39(6):461-470. doi: 10.1097/DBP.0000000000000575. PMID 29877990